CLINICAL TRIAL: NCT06750315
Title: CRP/ Albumin Ratio and Neutrophil Lymphocyte Ratio in Predicting Activity in IBD Patients
Brief Title: CRP /albumin Ratio and Neutrophil Lymphocyte Ratio in Predicting Activity in IBD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Ali Ahmed, Assistant Lecturer, Assiut University
Other Study IDs: CRP/ALB and N/L In active IBD
Record Dates: First submitted 2024-09-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: CRP/ALB ratio; N/L ratio
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aimed to assess the clinical utility of the NLR (neutrophil lymphocyte ratio) and CRP Albumin ratio in predicting activity of IBD Patients in assiut university

DETAILED DESCRIPTION:
IBD definition term for two conditions (Crohn's disease and ulcerative colitis) is a chronic idiopathic inflammatory disease affecting the large intestine. It is characterized by relapsing mucosal inflammation. The aim of treatment is to induce and maintain disease remission. Assessing disease activity may help in optimizing the management of IBD patients.

The neutrophil-to-lymphocyte ratio (NLR) is a simple index that can be calculated from the results of ordinary blood tests; it is calculated from a blood sample by dividing the absolute neutrophil count by the absolute lymphocyte count . As the NLR can reflect the systemic status of inflammation or immune response.

The underlying mechanism that the NLR was a predictor of clinilcal relapse in UC patients with Mucosal healing remains poorly understood. Neutrophils induce cytotoxicity and inflammation in UC. A high NLR value may be due to high activity in UC and lowered mucosal barrier function, which may lead to the migration of neutrophils through the gut microbiota .

CRP is routinely used as a surrogate measure of intestinal inflammation and as a prognostic measure of nonresponse to medical therapy and colectomy in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

Patients more than 18 years newly diagnosed as IBD

-

Exclusion Criteria:

* Patients Not DM Not cardiac failure Not Liver failure No malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pt more than 18 years not DM not cardiac failure Not Liver failure No malignancy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein /albumin ratio and neutrophil lymphocyte ratio in predicting activity in Inflammatory Bowel Disease Patients | 1 years
  Neutrophil lymphocyte ratio and CRP/Albumin ratio in detecting activity in IBD Patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University, Asyut
  - Assiut university hospital, Egypt, Assiut

REFERENCES:
- [Background] Torun S, Tunc BD, Suvak B, Yildiz H, Tas A, Sayilir A, Ozderin YO, Beyazit Y, Kayacetin E. Assessment of neutrophil-lymphocyte ratio in ulcerative colitis: a promising marker in predicting disease severity. Clin Res Hepatol Gastroenterol. 2012 Oct;36(5):491-7. doi: 10.1016/j.clinre.2012.06.004. Epub 2012 Jul 27. PMID 22841412
- [Background] Nguyen AL, Brick C, Liu D, Gibson DJ, Gibson PR, Sparrow MP. Clinical utility of C-reactive protein-to-albumin ratio in the management of patients with inflammatory bowel disease. JGH Open. 2024 Apr 15;8(4):e13059. doi: 10.1002/jgh3.13059. eCollection 2024 Apr. PMID 38623491
- [Background] Demir AK, Demirtas A, Kaya SU, Tastan I, Butun I, Sagcan M, Sahin S, Tasliyurt T, Yilmaz A. The relationship between the neutrophil-lymphocyte ratio and disease activity in patients with ulcerative colitis. Kaohsiung J Med Sci. 2015 Nov;31(11):585-90. doi: 10.1016/j.kjms.2015.10.001. Epub 2015 Oct 31. PMID 26678939
- [Background] Langley BO, Guedry SE, Goldenberg JZ, Hanes DA, Beardsley JA, Ryan JJ. Inflammatory Bowel Disease and Neutrophil-Lymphocyte Ratio: A Systematic Scoping Review. J Clin Med. 2021 Sep 17;10(18):4219. doi: 10.3390/jcm10184219. PMID 34575330